CLINICAL TRIAL: NCT05579327
Title: Withdrawal of Tiratricol Treatment in Males With Monocarboxylate Transporter 8 Deficiency (MCT8 Deficiency): A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Withdrawal of Tiratricol Treatment in Males With Monocarboxylate Transporter 8 Deficiency (MCT8 Deficiency)
Acronym: ReTRIACt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rare Thyroid Therapeutics International AB (Industry)
Collaborators: Premier Research (Other); Egetis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCT8-2021-3
Expanded Access: NCT05911399 (Available)
Record Dates: First submitted 2022-09-29; First posted 2022-10-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Monocarboxylate Transporter 8 Deficiency; Allan-Herndon-Dudley Syndrome
Keywords: MCT8; MCT8 deficiency; Allan-Herndon-Dudley syndrome; Tiratricol; Triac
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome | interventions — 3,3',5-triiodothyroacetic acid

STUDY DESIGN:
Intervention Model Description: Patients having demonstrated stable maintenance treatment with tiratricol will be randomized to receive placebo or tiratricol for 30 days or until reaching rescue criterion (serum total T3 > ULN of the participant's normal range, for a sample collected during the 30-day Randomized Treatment Period). In other words, the patients will be randomized to complete withdrawal of tiratricol treatment (placebo) for 30 days or to continue with the stable tiratricol maintenance treatment for 30 days. If during the 30 days, a rescue criterion (serum total T3 > ULN of the participant's normal range) is reached, the randomized treatment will be stopped, and the patient will go back on unblinded tiratricol treatment.
  Serum total T3 concentrations measured during the Randomized Treatment Period that are below the LLN of the normal range will not lead to any modifications to the blinded study drug administration schedule of daily tiratricol dosing.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tiratricol (Experimental)
  Interventions: Drug: Tiratricol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiratricol — Tiratricol tablets are flat tablets that contain 350 µg tiratricol. Treatment will be administered orally or via percutaneous endoscopic gastrostomy (PEG) tube; tablets will be suspended in water and, if needed, mixed with mashed food for oral administration or administered in water through the PEG tube as applicable.
  Arms: Tiratricol
Drug: Placebo — Placebo tablets will be identical in appearance to tiratricol tablets but contain no tiratricol. Treatment will be administered orally or via PEG tube; tablets will be suspended in water and, if needed, mixed with mashed food for oral administration or administered in water through the PEG tube as applicable. During the Randomized Treatment Period, participants will receive the same number of tablets as the stable dose of open-label tiratricol they were receiving before randomization.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized phase 3 multicenter placebo-controlled study in at least 16 evaluable male participants diagnosed with MCT8 deficiency. Male participants, from 4 years of age (at randomization) and having demonstrated stable maintenance treatment with tiratricol, will be randomized to receive placebo or tiratricol for 30 days or until reaching rescue criterion (serum total triiodothyronine [T3] > upper limit of normal [ULN] of the participant's normal range, for a sample collected during the 30-day Randomized Treatment Period). The research hypothesis to be tested is that, for participants in the placebo group, removal of tiratricol will lead to an increase of serum total T3 concentration, measured by liquid chromatography with tandem mass spectrometry (LC/MS/MS), above the ULN and requirement of rescue treatment with tiratricol, compared to those who continue to receive tiratricol.

DETAILED DESCRIPTION:
The Screening Period includes a Screening Visit and a period of open-label treatment in which a stable maintenance dose of tiratricol, essential for progression into the Randomized Treatment Period, will be established. The duration of this period will vary depending on whether the participant is currently receiving treatment with tiratricol at the time of enrollment in the study (Cohort A), or if they are considered to be tiratricol treatment-naïve (Cohort B). Participants are considered to be tiratricol-naïve if they have never previously been administered tiratricol, or have previously received tiratricol but are not receiving tiratricol at the time of enrollment.

For participants in Cohort A, once eligibility is confirmed during the Screening Visit, the study starts with a Run-in Period to ensure that participants are being administered a stable dose of tiratricol, as determined by meeting the Stable Dose Criterion.

For participants in Cohort B, once eligibility is confirmed during the Screening Visit, the study starts with a Dose Titration Period to allow titration to a stable dose of tiratricol, as determined by meeting the Stable Dose Criterion.

The Stable Dose Criterion is defined as at least 4 weeks' treatment (during the period from the start of screening to randomization) at a fixed daily dose that is targeting a serum total T3, measured by LC/MS/MS, at the lower limit of normal (LLN) with at least 2 consecutive serum total T3 results that are within the study titration range: within 20% below the LLN to the 75th percentile of the normal range for serum total T3 (i.e., LLN + 0.75×[ULN-LLN]).

An evaluable participant is defined as a participant who completes the Randomized Treatment Period either by completing 30 days of double-blind treatment without meeting the rescue criterion or by meeting the rescue criterion.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants diagnosed with a pathogenic mutation in the MCT8 gene, confirmed with a genetic test.
2. Serum total T3 concentration above the ULN of the age specific normal range:

   1. at the time of diagnosis (or the closest sample taken prior to first ever treatment with tiratricol) for participants who are currently treated with tiratricol
   2. in the Screening Visit sample, or most recent standard of care sample prior to screening, for participants who have never received and/or currently not receiving tiratricol.
3. Participants will be aged 4 years or older at the time of randomization. Participants entering screening who are <4 years of age but expected to be aged 4 years at randomization should be discussed with the medical monitor.
4. Signed and dated informed consent form from the parents or legal guardian.

Exclusion Criteria:

1. Major illness or recent major surgery unrelated to MCT8 deficiency (in the principal investigator's judgement), defined as:

   * Conditions requiring repeated hospitalizations that are likely to confound ability to participate in the trial.
   * Major illness in the 3 months prior to the screening visit that is likely to confound the ability of the participant to participate fully within the trial and/or confound the assessment of serum total T3 and/or safety.
   * Major surgery within the 3 months prior to the screening visit or planned to take place during the study, including but not limited to major abdominal/thoracic/neurosurgical procedures.
   * Major/minor abdominal and/or maxillofacial surgery that may inhibit the administration and/or absorption of study drug.
2. Body weight <10 kg at the Screening Visit.
3. Patients who are participating, or intend to participate, in other therapeutic and/or interventional clinical studies during the study period.
4. History of allergic reactions to components of tiratricol or any excipients in the investigational product (IP).
5. Participants with any contra-indication for treatment with tiratricol or any excipients in the IP.
6. Participants using other T3 analogues, levothyroxine, or propylthiouracil.

Randomization Criteria:

In addition to the eligibility criteria, participants must meet further criteria at the time of randomization to enter the Randomized Treatment Period.

1. Confirmation that the "Stable Dose Criterion" has been met.
2. Absence of any new or exacerbated medical or surgical condition that fulfils Exclusion criterion #1.
3. Confirmation that participant is at least 4 years of age at the time of randomization.

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Rate of change from baseline in serum total T3 during the 30-day double blind Randomized Treatment Period. | During the 30-day double blind Randomized Treatment Period.
Proportion of participants who meet the rescue criterion (serum total T3 > ULN) during the 30-day double-blind Randomized Treatment Period. | During the 30-day double-blind Randomized Treatment Period.

SECONDARY OUTCOMES:
Change in serum thyroid hormone variables (T3, T4, TSH, fT3, and fT4). | From i) baseline to the end of Randomized Treatment Period, ii) screening to End of Study, iii) initiation of tiratricol administration at enrolment to the last measurement prior to randomization.
Change in clinical endpoints: Heart Rate, Systolic Blood Pressure and Rate Pressure Product (heart rate × systolic blood pressure). | From i) baseline to the end of Randomized Treatment Period, ii) initiation of tiratricol administration at screening to the last measurement prior to randomization.
Change in clinical endpoints: Heart Rate, Systolic Blood Pressure, Rate Pressure Product (heart rate × systolic blood pressure) and body weight. | From Screening to End of Study.
Safety endpoints: Adverse events, Safety laboratory variables, Standard vital signs variables, Weight, ECG evaluations and Physical examinations. | From the start of the Run-in/Dose Titration Period to the end of study.
  Safety laboratory variables (full blood count, serum renal and liver biomarkers, total and LDL cholesterol), Standard vital signs variables (temperature, respiratory rate, pulse rate and blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Bauer, MD, Principal Investigator — Children's Hospital of Philadelphia; W. E. Visser, MD, Principal Investigator — Erasmus Medical Center
Locations (8):
- United States (6):
  - Rare Disease Research, LLC, Kissimmee, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Rare Disease Research, LLC, Hillsborough, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Tranquil Clinical and Research Consulting Services, Webster, Texas
- Erasmus MC, Rotterdam, Netherlands
- Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided